CLINICAL TRIAL: NCT05827120
Title: Long-term Effect of Different Modes of Endovascular Therapy in Combination With Anticoagulation Treatment in Patients With Acute Extensive Deep Vein Thrombosis (LEVANTE Research)
Brief Title: Endovascular Therapy in Patients With Acute Deep Vein Thrombosis
Acronym: LEVANTE
Status: Completed | Type: Observational
Sponsor: National Institute of Cardiovascular Diseases, Slovakia (Other)
Collaborators: East Slovakia Institute of Cardiovascular Diseases in Košice, Slovakia (Unknown); Central Slovakia Institute of Cardiovascular Diseases in Banská Bystrica, Slovakia (Unknown)
Responsible Party: Principal Investigator, Juraj Maďarič, MD, assoc. prof. Juraj Maďarič, PhD., MPH, Department of Cardiology and Angiology - head of the unit, National Institute of Cardiovascular Diseases, Slovakia
Other Study IDs: 65176743 / LEVA002NUSCH
Record Dates: First submitted 2023-04-06; First posted 2023-04-24 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Acute Deep Venous Thrombosis
Keywords: deep venous thrombosis; endovascular thrombectomy; anticoagulation
MeSH Terms: conditions — Venous Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Thrombectomy plus local thrombolysis group: Thrombectomy plus local thrombolysis group - patients treated by mechanical thrombectomy mostly followed by catheter directed thrombolysis (CDT), or by pharmaco-mechanical thrombectomy (PMT) - combination of some form of mechanical disruption of the thrombus in conjunction with chemical lysis. Thrombolysis by alteplase 1mg/hour. Procedure followed by anticoagulation therapy.
  Interventions: Device: Mechanical / pharmacomechanical thrombectomy plus local catheter directed thrombolysis
- Local catheter directed thrombolysis alone group: Local catheter directed thrombolysis alone group - patients treated by dedicated catheter for local thrombolysis with side holes placed across the acute thrombus - continuous infusion of alteplase 1mg per hour simultaneously with unfractionated heparine in anticoagulation dosage. Without mechanical or pharmaco-mechanical thrombectomy. Procedure followed by anticoagulation therapy.
  Interventions: Device: Local catheter directed thrombolysis alone

INTERVENTIONS:
Device: Mechanical / pharmacomechanical thrombectomy plus local catheter directed thrombolysis — * Catheter directed thrombolysis (CDT): dedicated thrombolytic catheter with side holes is placed across the acute thrombus, and slow, continuous infusion (through the catheter, or both through the catheter and sheath) of a chemical thrombolysis agent is applied - alteplase 1mg/hour plus unfractionated heparine in anticoagulation dosage;
  * Mechanical thrombectomy: mechanical aspiration of fresh thrombus;
  * Pharmacomechanical thrombectomy (PMT): combination of mechanical disruption of the thrombus, and its aspiration, with simultaneous application of alteplase via dedicated catheter - instilation of acute/subacute thrombus with its subsequent aspiration;
  Groups: Thrombectomy plus local thrombolysis group
Device: Local catheter directed thrombolysis alone — - Catheter directed thrombolysis (CDT): dedicated thrombolytic catheter with side holes is placed across the acute thrombus, and slow, continuous infusion (through the catheter, or both through the catheter and sheath) of a chemical thrombolysis agent is applied - alteplase 1mg/hour plus unfractionated heparine in anticoagulation dosage;
  Groups: Local catheter directed thrombolysis alone group

SUMMARY:
Despite optimal anticoagulation therapy of patients with proximal deep vein thrombosis (DVT), there is still high number of patients suffering from post-thrombotic syndrome (PTS) due to the chronic venous occlusion, suboptimal collateralization, and venous valvular dysfunction. Last two decades endovascular catheter-based treatment modalities have been tested and used in an attempt to reduce incidence and symptoms of PTS in selected patients.

Especially, patients with extensive iliofemoral DVT have an increased risk of PTS. In an effort to accelerate thrombus dissolution or thrombus extraction, the endovascular removal of acute venous thrombus has been introduced as therapeutic option in patients with extensive iliofemoral DVT.

Randomized trials of catheter-based strategies for thrombus removal have documented improved vein patency, preserved valves function, and reduced post-thrombotic syndrome.

The aim of our study is to evaluate the safety and efficacy of different types of endovascular methods of treatment followed by anticoagulation therapy in patients with acute extensive DVT. Retrospective multicentre analysis of app 100 patients scheduled for endovascular treatment of extensive DVT. The results of mechanical/pharmacomechanical thrombectomy followed by local catheter directed thrombolysis (CDT), will be compared with CDT alone, or with ultrasound-accelerated thrombolysis. The 24-month incidence of PTS assessed by Villalta scoring system, major bleeding complications, the rate of venous recanalization, recurrence of DVT, and other end-points will be evaluated.

DETAILED DESCRIPTION:
Aim: The aim of the study is to evaluate the long-term incidence of PTS in patients treated by different endovascular methods and protocols in combination with anticoagulation medication in patients with acute extensive DVT.

Hypothesis: Mechanical / pharmacomechanical thrombectomy (PMT) following by CDT and further anticoagulation therapy is safe and effective mode of acute DVT treatment with reduction of PTS after 24 months in comparison with historical data and with other modes of endovascular therapy.

Methods: Retrospective multicentre analysis of patients scheduled to interventional endovenous treatment of extensive DVT.

The major end-point:

1. The development of PTS during the 24-month follow-up period

The minor end-points:

1. The occurrence of major bleeding and live-threatening bleeding episodes
2. The development of PTS during the 6-month and 12-month follow-up period
3. The rate of venous recanalization after intervention assessed by ultrasound
4. The occurrence of pulmonary embolism
5. Recurrence of DVT
6. Mortality, myocardial infarction, stroke during follow-up

The occurrence of PTS will be assessed by clinical evaluation and by Villalta scoring system.

Patients suitable for endovascular therapy and for enrolment into study:

* first episode of acute iliofemoral DVT
* duration of symptoms <14 days
* symptomatic patients with no or limited response to initial anticoagulation therapy in terms of symptomatology and signs of recanalization
* low bleeding risk
* good functional capacity and life expectancy

Endovascular procedures retrospectively analysed:

* Catheter directed thrombolysis (CDT): dedicated infusion catheter with side holes is placed across the acute thrombus, and slow, continuous infusion (through the catheter, or both through the catheter and sheath) of a chemical thrombolysis agent is initiated (alteplase 1mg per hour simultaneously with unfractionated heparine (UFH) in anticoagulation dosage); activated partial thromboplastin time (APTT), fibrinogen (Fbg), and blood count must be controlled;
* Mechanical thrombectomy: mechanical aspiration of fresh thrombus; mostly followed by CDT;
* Pharmacomechanical thrombectomy (PMT): combination of some form of mechanical disruption of the thrombus in conjunction with chemical lysis. There is evidence that PMT quickens thrombolysis compared with CDT alone. Dedicated devices combining chemical thrombolysis via power-pulse fluid plus plasminogen activator thrombus penetration, with rheolytic fluid-based disruption of thrombus and catheter-based aspiration thrombectomy.
* Ultrasound-accelerated thrombolysis combines chemical CDT with low-power high-frequency ultrasound application to the proprietary infusion catheter/wire combination, with the ultrasonic vibration purported to hasten thrombus disruption; the addition of ultrasound during lytic infusion increases the surface area of the fibrin, thereby permitting more efficient binding of the plasminogen activator to the fibrin-bound plasminogen
* Stenting of residual thrombotic lesions, and stenting of common iliac vein compression in the presence of May-Thurner syndrome;

Peri-procedure and post-procedure care retrospectively analysed:

* continuous in-hospital monitoring to minimize CDT-related complications;
* APTT, Fbg concentration, and blood count are monitored;
* Anticoagulation after endovascular procedure as standard regimen, if no contraindications, mostly during the 6-month time period; longer anticoagulation regimen is at discretion of treated centre and physician;
* after venous stenting may be consider clopidogrel along with anticoagulation therapy for 1 month (not proven); Ultrasound evaluation during follow-up (data from documentation)
* recanalization - no residual thrombosis
* recanalization >50%
* recanalization <50%
* minimal US signs of recanalization/no recanalization Post-thrombotic syndrome: clinical evaluation and/or Villalta score
* No PTS: Villalta <5 points
* Mild: 5-9 points
* Moderate: 10-14 points
* Severe PTS: ≥15 points/venous ulcer

ELIGIBILITY:
Inclusion Criteria:

* first episode of acute iliofemoral DVT
* duration of symptoms <14 days
* symptomatic patients with no or limited response to initial anticoagulation therapy in terms of symptomatology and signs of recanalization
* low bleeding risk
* good functional capacity and life expectancy

Exclusion Criteria:

* - presence of malignity (2 centers out of 3)
* pregnancy
* haemorrhagic diathesis / high risk of bleeding
* negative prognosis of survival
* renal / hepatic failure
* chronic course of DVT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for endovascular treatment of extensive deep venous thrombosis (DVT)
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2021-03-23 (Actual); Primary Completion 2023-02-24 (Actual); Study Completion 2023-02-24 (Actual)

PRIMARY OUTCOMES:
Post-thrombotic syndrome | 24-month follow-up period
  The occurrence of PTS will be assessed by clinical evaluation and by Villalta scoring system (0-33), higher scores mean a worse outcome.

SECONDARY OUTCOMES:
The occurrence of major bleeding and live-threatening bleeding episodes | periprocedural, in-hospital (up to day 7), 24 months
  clinical and laboratory evaluation of bleeding
The development of PTS during the 6-month and 12-month follow-up period | 6-month and 12-month follow-up period
  The occurrence of PTS will be assessed by clinical evaluation and by Villalta scoring system (0-33), higher scores mean a worse outcome.
The rate of venous recanalization after intervention | early - in-hospital (up to day 7), 6-month
  assessed by ultrasound
The occurrence of pulmonary embolism | early - in-hospital (up to day 7), 12-month, 24-month follow-up
  clinical evaluation
Recurrence of DVT | 12-month, 24-month follow-up
  clinical and ultrasound evaluation
Mortality, MI, stroke during follow-up | In-hospital (up to day 7), 12-month, 24-month follow-up
  history assessment

CONTACTS AND LOCATIONS:
Overall Officials: Juraj Maďarič, assoc. prof, Principal Investigator — National Institute of Cardiovascular Diseases
Locations (3):
- Slovakia (3):
  - Central Slovakia Institute of Cardiovascular Diseases in Banská Bystrica, Banská Bystrica
  - National Institute of Cardiovascular Diseases, Slovakia, Bratislava
  - East Slovakia Institute of Cardiovascular Diseases in Košice, Košice

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kahn SR, Comerota AJ, Cushman M, Evans NS, Ginsberg JS, Goldenberg NA, Gupta DK, Prandoni P, Vedantham S, Walsh ME, Weitz JI; American Heart Association Council on Peripheral Vascular Disease, Council on Clinical Cardiology, and Council on Cardiovascular and Stroke Nursing. The postthrombotic syndrome: evidence-based prevention, diagnosis, and treatment strategies: a scientific statement from the American Heart Association. Circulation. 2014 Oct 28;130(18):1636-61. doi: 10.1161/CIR.0000000000000130. Epub 2014 Sep 22. No abstract available. PMID 25246013
- [Background] Razavi MK, Jaff MR, Miller LE. Safety and Effectiveness of Stent Placement for Iliofemoral Venous Outflow Obstruction: Systematic Review and Meta-Analysis. Circ Cardiovasc Interv. 2015 Oct;8(10):e002772. doi: 10.1161/CIRCINTERVENTIONS.115.002772. PMID 26438686
- [Background] Comerota AJ, Grewal N, Martinez JT, Chen JT, Disalle R, Andrews L, Sepanski D, Assi Z. Postthrombotic morbidity correlates with residual thrombus following catheter-directed thrombolysis for iliofemoral deep vein thrombosis. J Vasc Surg. 2012 Mar;55(3):768-73. doi: 10.1016/j.jvs.2011.10.032. Epub 2012 Jan 24. PMID 22277690
- [Background] Tick LW, Doggen CJ, Rosendaal FR, Faber WR, Bousema MT, Mackaay AJ, VAN Balen P, Kramer MH. Predictors of the post-thrombotic syndrome with non-invasive venous examinations in patients 6 weeks after a first episode of deep vein thrombosis. J Thromb Haemost. 2010 Dec;8(12):2685-92. doi: 10.1111/j.1538-7836.2010.04065.x. PMID 20860679
- [Background] Delis KT, Bountouroglou D, Mansfield AO. Venous claudication in iliofemoral thrombosis: long-term effects on venous hemodynamics, clinical status, and quality of life. Ann Surg. 2004 Jan;239(1):118-26. doi: 10.1097/01.sla.0000103067.10695.74. PMID 14685109
- [Background] Kearon C, Akl EA, Ornelas J, Blaivas A, Jimenez D, Bounameaux H, Huisman M, King CS, Morris TA, Sood N, Stevens SM, Vintch JRE, Wells P, Woller SC, Moores L. Antithrombotic Therapy for VTE Disease: CHEST Guideline and Expert Panel Report. Chest. 2016 Feb;149(2):315-352. doi: 10.1016/j.chest.2015.11.026. Epub 2016 Jan 7. PMID 26867832
- [Background] Jaff MR, McMurtry MS, Archer SL, Cushman M, Goldenberg N, Goldhaber SZ, Jenkins JS, Kline JA, Michaels AD, Thistlethwaite P, Vedantham S, White RJ, Zierler BK; American Heart Association Council on Cardiopulmonary, Critical Care, Perioperative and Resuscitation; American Heart Association Council on Peripheral Vascular Disease; American Heart Association Council on Arteriosclerosis, Thrombosis and Vascular Biology. Management of massive and submassive pulmonary embolism, iliofemoral deep vein thrombosis, and chronic thromboembolic pulmonary hypertension: a scientific statement from the American Heart Association. Circulation. 2011 Apr 26;123(16):1788-830. doi: 10.1161/CIR.0b013e318214914f. Epub 2011 Mar 21. PMID 21422387
- [Background] Meissner MH, Gloviczki P, Comerota AJ, Dalsing MC, Eklof BG, Gillespie DL, Lohr JM, McLafferty RB, Murad MH, Padberg F, Pappas P, Raffetto JD, Wakefield TW; Society for Vascular Surgery; American Venous Forum. Early thrombus removal strategies for acute deep venous thrombosis: clinical practice guidelines of the Society for Vascular Surgery and the American Venous Forum. J Vasc Surg. 2012 May;55(5):1449-62. doi: 10.1016/j.jvs.2011.12.081. Epub 2012 Apr 1. PMID 22469503
- [Background] Sharifi M, Bay C, Mehdipour M, Sharifi J; TORPEDO Investigators. Thrombus Obliteration by Rapid Percutaneous Endovenous Intervention in Deep Venous Occlusion (TORPEDO) trial: midterm results. J Endovasc Ther. 2012 Apr;19(2):273-80. doi: 10.1583/11-3674MR.1. PMID 22545895
- [Background] Kahn SR, Julian JA, Kearon C, Gu CS, Cohen DJ, Magnuson EA, Comerota AJ, Goldhaber SZ, Jaff MR, Razavi MK, Kindzelski AL, Schneider JR, Kim P, Chaer R, Sista AK, McLafferty RB, Kaufman JA, Wible BC, Blinder M, Vedantham S; ATTRACT Trial Investigators. Quality of life after pharmacomechanical catheter-directed thrombolysis for proximal deep venous thrombosis. J Vasc Surg Venous Lymphat Disord. 2020 Jan;8(1):8-23.e18. doi: 10.1016/j.jvsv.2019.03.023. PMID 31843251
- [Background] Comerota AJ, Kearon C, Gu CS, Julian JA, Goldhaber SZ, Kahn SR, Jaff MR, Razavi MK, Kindzelski AL, Bashir R, Patel P, Sharafuddin M, Sichlau MJ, Saad WE, Assi Z, Hofmann LV, Kennedy M, Vedantham S; ATTRACT Trial Investigators. Endovascular Thrombus Removal for Acute Iliofemoral Deep Vein Thrombosis. Circulation. 2019 Feb 26;139(9):1162-1173. doi: 10.1161/CIRCULATIONAHA.118.037425. PMID 30586751
- [Background] Lu T, Loh TM, El-Sayed HF, Davies MG. Single-center retrospective review of ultrasound-accelerated versus traditional catheter-directed thrombolysis for acute lower extremity deep venous thrombosis. Vascular. 2017 Oct;25(5):525-532. doi: 10.1177/1708538117702061. Epub 2017 Apr 3. PMID 28372484
- [Background] Prandoni P, Kahn SR. Post-thrombotic syndrome: prevalence, prognostication and need for progress. Br J Haematol. 2009 May;145(3):286-95. doi: 10.1111/j.1365-2141.2009.07601.x. Epub 2009 Feb 13. PMID 19222476
- [Background] Haig Y, Enden T, Grotta O, Klow NE, Slagsvold CE, Ghanima W, Sandvik L, Hafsahl G, Holme PA, Holmen LO, Njaaastad AM, Sandbaek G, Sandset PM; CaVenT Study Group. Post-thrombotic syndrome after catheter-directed thrombolysis for deep vein thrombosis (CaVenT): 5-year follow-up results of an open-label, randomised controlled trial. Lancet Haematol. 2016 Feb;3(2):e64-71. doi: 10.1016/S2352-3026(15)00248-3. Epub 2016 Jan 6. PMID 26853645
- [Background] Vedantham S, Goldhaber SZ, Julian JA, Kahn SR, Jaff MR, Cohen DJ, Magnuson E, Razavi MK, Comerota AJ, Gornik HL, Murphy TP, Lewis L, Duncan JR, Nieters P, Derfler MC, Filion M, Gu CS, Kee S, Schneider J, Saad N, Blinder M, Moll S, Sacks D, Lin J, Rundback J, Garcia M, Razdan R, VanderWoude E, Marques V, Kearon C; ATTRACT Trial Investigators. Pharmacomechanical Catheter-Directed Thrombolysis for Deep-Vein Thrombosis. N Engl J Med. 2017 Dec 7;377(23):2240-2252. doi: 10.1056/NEJMoa1615066. PMID 29211671
- [Background] Leung DA, Blitz LR, Nelson T, Amin A, Soukas PA, Nanjundappa A, Garcia MJ, Lookstein R, Simoni EJ. Rheolytic Pharmacomechanical Thrombectomy for the Management of Acute Limb Ischemia: Results From the PEARL Registry. J Endovasc Ther. 2015 Aug;22(4):546-57. doi: 10.1177/1526602815592849. Epub 2015 Jun 24. PMID 26109628